CLINICAL TRIAL: NCT03442153
Title: Comparative Efficacy and Tolerability of No7 in Osteoarthritis of the Knee: A Double Blind, Randomized, Placebo Controlled Clinical Study
Brief Title: Comparative Efficacy and Tolerability of No7 in Osteoarthritis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ambrosia - SupHerb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ambrosia
Record Dates: First submitted 2018-01-09; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The product in not drug or medical device (but a dietary supplement). There are 76 participants divided inti 2 groups : experimental group (38) and Placebo group (38). The period of the intervention: 90 days
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solgar No7 (Experimental): Aflapin 100 mg and Collagen UC2 40 mg by mouth every 24 hours for 90 days
  Interventions: Dietary Supplement: Solgar No7 Complex
- Placebo for Solgar No7 (Placebo Comparator): Placebo 1 Capsule by mouth, every 24 hours for 90 days
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Solgar No7 Complex — Solgar No7 Capsules
  Arms: Solgar No7
Dietary Supplement: placebo — Placebo tablets Cellulose
  Other Names: Placebo for Solgar No7
  Arms: Placebo for Solgar No7

SUMMARY:
This study evaluates the effect of dietary supplement Solgar No7 in 76 adult Osteoarthritis of the Knee Patients, while the other half will receive placebo.

DETAILED DESCRIPTION:
Solgar No7 is a Dietary Supplement marketed in Israel on a regular basis with the approval of the Israeli Ministry of Health. The product is based on Herbal Extracts and Vitamins. The individual components of the product were effective in some studies in relieving pain and inflammation in such patients. This Study evaluates the effect of these components as a complex.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis (at least 2-nd grade according to Kellgren Classification)
* Ability to walk independently
* Pain Intensity of 4 or more according to Visual Analogue Scale
* NSAIDs usage of 5 times or more per month during 3 months before the intervention
* Ability to understand the benefits and risks of the proposed treatment and can provide answers to the required questions and fill out a questionnaire in Hebrew
* Early consent of participants not to start a new treatment for Osteoarthritis including medication, surgery, physiotherapy, laser therapy, etc. during the period of the study (3 months) - except for a clear medical need (should report to the investigators immediately)

Exclusion Criteria:

* Inflammatory Arthropathy, Severe Rheumatoid Arthritis, Psoriatic Arthritis or Gout
* History of injection of pharmacological material (steroids, anesthetic, hyaluronic acid or any other pharmacological substance) into the knee joint during the six months prior to the start of the study
* Taking of biological drugs that may affect inflammatory conditions (such as anti-TNF- alpha, etc.) or oral PO steroids - even if given to another disease, for more than 5 days during 3 months prior to the start of the study
* Chronic administration of any anti-inflammatory drug during the study period and / or at least one month prior to commencement of the study.
* Chronic administration of medical cannabis
* Use of analgetics in a formulation that provides a half-life of over 24 hours (eg, Butrans, Fentanyl)
* Chronic use of vitamin K antagonists, Heparin, Enoxaparin
* Injury to the knee during six months prior to the experiment
* Expectations of surgical intervention, physiotherapy or other treatment of osteoarthritis before the end of the study period
* Significant irregularities in renal or liver function, active malignant disease in the last 3 years, heart failure, uncontrolled hypertension, active peptic ulcer, hematologic diseases, severe neurological diseases, and mental illness with seizures in the last two years.
* Peripheral neuropathy that treated by any drug
* High alcohol consumption (over 2 standard doses per day)
* Sensitivity to one of the ingredients and / or sensitivity to NSAIDs. It is Possible to include a patient who is sensitive to a specific drug from the family of NSAIDs, but can take other drugs from this family.
* Any medical condition or treatment which, in the opinion of the investigators, may mask the results of the study and / or interfere with the research questions and / or terminate the research properly and / or endanger the participant in any way during the course of the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity Reported to the Doctor after one month of the treatment. Each item is scored 0-10 (0=no pain; 10=pain as bad as can be), yielding a total between 0 and 30.
  Self reported pain intensity in the scale 1-10

SECONDARY OUTCOMES:
Knee Stiffness | nee Stiffness checked by the Doctor after one month of treatment. Each item is scored 0-10 (0=no pain; 10=pain as bad as can be), yielding a total between 0 and 30
  The stiffness of the knee according to the doctor evaluation
Non Steroidal Anti Inflammatory Drugs Usage | Pain Medication Usage as Reported to the Doctor after one month of treatment. Each item is scored as a number of the dose units that were used during the all period (0=no medications, 1=only one dose of medication etc)
  Self reported Non Steroidal Anti Inflammatory Drugs Usage
Adverse Reactions | Adverse Reactions as Reported to the Doctor over the period of the treatment. Each item is scored as a number of the dose units that were used during the all period (0=no adverse reactions, 1=only one adverse reaction etc)
  Self reported Adverse Reactions

CONTACTS AND LOCATIONS:
Overall Officials: Guy Rubin, Principal Investigator — HaEmek Medical Center, Israel

IPD SHARING:
Plan to Share IPD: No